CLINICAL TRIAL: NCT04679831
Title: Clinical Evaluation of Ujiplus®, a Porridge Snack With Deworming Properties for Activity Against Schistosoma Mansoni
Brief Title: Clinical Evaluation of Ujiplus® Against Schistosoma Mansoni
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: Kanazawa University (Other)
Responsible Party: Principal Investigator, Elijah M. Songok, Proffesor, Kenya Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSC2580/2
Record Dates: First submitted 2020-12-18; First posted 2020-12-22 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Schistosoma Mansoni
MeSH Terms: conditions — Schistosomiasis | interventions — Praziquantel

STUDY DESIGN:
Intervention Model Description: Dietary Supplement: Ujiplus Ujiplus flour, a nutritional supplement. The flour will be used to prepare porridge and each child is given a serving of 300 ml every school day for 90 days.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ujiplus® porridge (Experimental): Arm receiving porridge fortified with dried papaya seeds (Ujiplus)
  Interventions: Dietary Supplement: Ujiplus®
- Praziquantel 400mg (Active Comparator): Arm receiving the approved Praziquantel treatment of 400mg once with plain porridge daily (without papaya seeds)
  Interventions: Drug: Praziquantel 400mg

INTERVENTIONS:
Dietary Supplement: Ujiplus® — Ujiplus® flour, a nutritional supplement will be used to prepare porridge, and each child will be given a serving of 300 ml every school day for 90 days.
  Arms: Ujiplus® porridge
Drug: Praziquantel 400mg — 400mg of Praziquantel will be given to each child once at the beginning of the study and maize flour porridge fortified only with micronutrients cooked and served to each child, 300 ml per every school day for 90 days,
  Other Names: Biltricide
  Arms: Praziquantel 400mg

SUMMARY:
Schistosomiasis is classified as among the world's neglected tropical diseases (NTD). Morbidity due to Schistosoma mansoni (S. mansoni) is greatest among school-age children who typically have the highest burden of infection. In 2001, World Health Organization (WHO) passed a resolution for large-scale mass drug administration (MDA) using chemotherapy to deworm vulnerable children through school-based programs. While MDA has significantly contributed to reducing the burden of these infections, several concerns still exist over the large-scale use of chemotherapeutic drugs in deworming. The large population of children and the high frequency of dosage may pose a challenge to the sustainability of these programs. Further, the MDAs exert increasing drug pressure on parasite populations, a circumstance that is likely to favor parasite genotypes that can resist chemotherapy. Additionally, the current school-based MDA does not consider child malnutrition a very common malady in African countries. The greatest shortcoming is that currently approved S. mansoni chemotherapeutic treatment, Praziquantel is not recommended for children under six years of age due to its perceived toxicity. This excludes a highly vulnerable group from treatment.

The above has called for alternative management options for S. mansoni among school and pre-school age children. The current study seeks to test the feasibility of the use of a nutritional supplement (Ujiplus®), as a potential deworming strategy against S. mansoni. Ujiplus® is a porridge flour fortified with papaya (Carica papaya) seeds extracts. In a previous study (NCT 027-25255), the product was found to have an effect on soil-transmitted helminths among a group of school children with no serious adverse events. We intend to evaluate the efficacy of Ujiplus® when given through school feeding programs and compare the outcome with praziquantel- the recommended MDA agent for deworming school children. The investigators will design and formulate the Ujiplus®, and test it among children in four primary schools in Mbita, Homabay county, Kenya.

DETAILED DESCRIPTION:
Background: Schistosomiasis is classified as among the world's neglected tropical diseases (NTD). Morbidity due to Schistosoma mansoni (S.mansoni) is greatest among school-age children who typically have the highest burden of infection. In 2001, World Health Organization (WHO) passed a resolution for large-scale mass drug administration (MDA) using chemotherapy to deworm vulnerable children through school-based programs. While MDA has significantly contributed to reducing the burden of these infections, several concerns still exist over the large-scale use of chemotherapeutic drugs in deworming. The large population of children and the high frequency of dosage may pose a challenge to the sustainability of these programs. Further, the MDAs exert increasing drug pressure on parasite populations, a circumstance that is likely to favor parasite genotypes that can resist chemotherapy. Moreover, chemotherapeutic drugs are not recommended for children under the age of 6 years due to their toxicity, despite the fact that this is the age group most infected with S. mansoni. Additionally, the current school-based MDA does not consider child malnutrition a very common malady in African countries.

Based on the above, we have designed a nutritional food supplement, Ujiplus®, with the potential as a homegrown mass drug administration tool against intestinal parasites including S.mansoni. Porridge (Uji) made from corn flour is one of the most prevalent traditional school meal snacks in developing countries. Because of its low cost, and popularity in schools, it has been adopted as a component in school meals, often prepared and given as a snack at break time. To enhance its effect, we have fortified the Uji flour with micronutrients and extracts from papaya (Carica papaya) seeds to form Ujiplus®. Carica papaya seeds have been found in various studies to have an anthelminthic effect with benzyl isothiocyanate (BITC) as the potential active ingredient. In a previous clinical trial, Ujiplus® reduced the Ascaris lumbricoides egg count by 63.9% after the two month period as compared to the albendazole arm, 78.8%.

In this study, primary school children (ages 6-8) from four schools in Homabay County Kenya will be randomized into two arms: Children from two schools will receive 300 ml Ujiplus® porridge daily (test school), and the other two schools will receive a similar serving of plain porridge (cornflour and micronutrients only) with Praziquantel. Prior to the randomization, an initial baseline stool microscopy analysis will be done to determine the presence and intensity of intestinal worms. Core indicators of nutrition-height, weight, and hemoglobin counts-will also be assessed. The children will be monitored daily for three months and final stool sample analysis and clinical monitoring done at the end of the study. Baseline and follow-up data will be collected through Redcap software (Vanderbilt, Nashville, Tenn) analyzed and compared through the latest software of SAS statistical package.

ELIGIBILITY:
Inclusion Criteria:

* Consenting parents and guardians

Exclusion Criteria:

* Children with known allergy to papaya fruit products

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Parasite egg count | 90 days after randomization
  Parasitic eggs in a stool sample will be counted at the end of the intervention, using the Katz thick smear technique, and recorded as eggs per gram of faeces (EPG)

SECONDARY OUTCOMES:
Body Mass Index for age | 90 days after intervention
  Height, Weight and age will be collected. BMI will be calculated using WHO guidelines.
Class attendance | 90 days after randomization
  The class register used by the class teacher to record daily student attendance will be used to gather information on attendance, enrollment, and retention of students.
Haemoglobin levels | 90 days after randomization
  Blood sample will be taken for hemoglobin amounts at start and end of intervention
Number of children with Schistosoma mansoni | 90 days after randomization
  Number of children with Schistosoma mansoni will be recorded at start and end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elijah M Songok, PhD, Principal Investigator — Kenya Medical Research Institute
Locations (1):
- Mbita, Mbita, Kenya

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting September 2021
Access Criteria: Publication

REFERENCES:
- [Background] Avila S, Kugo M, Silveira Hornung P, Apea-Bah FB, Songok EM, Beta T. Carica papaya seed enhances phytochemicals and functional properties in cornmeal porridges. Food Chem. 2020 Sep 1;323:126808. doi: 10.1016/j.foodchem.2020.126808. Epub 2020 Apr 15. PMID 32335458
- [Background] Kugo M, Keter L, Maiyo A, Kinyua J, Ndemwa P, Maina G, Otieno P, Songok EM. Fortification of Carica papaya fruit seeds to school meal snacks may aid Africa mass deworming programs: a preliminary survey. BMC Complement Altern Med. 2018 Dec 7;18(1):327. doi: 10.1186/s12906-018-2379-2. PMID 30526582
- [Background] Okeniyi JA, Ogunlesi TA, Oyelami OA, Adeyemi LA. Effectiveness of dried Carica papaya seeds against human intestinal parasitosis: a pilot study. J Med Food. 2007 Mar;10(1):194-6. doi: 10.1089/jmf.2005.065. PMID 17472487
- [Background] Kermanshai R, McCarry BE, Rosenfeld J, Summers PS, Weretilnyk EA, Sorger GJ. Benzyl isothiocyanate is the chief or sole anthelmintic in papaya seed extracts. Phytochemistry. 2001 Jun;57(3):427-35. doi: 10.1016/s0031-9422(01)00077-2. PMID 11393524
- [Background] Sapaat A, Satrija F, Mahsol HH, Ahmad AH. Anthelmintic activity of papaya seeds on Hymenolepis diminuta infections in rats. Trop Biomed. 2012 Dec;29(4):508-12. PMID 23202594